CLINICAL TRIAL: NCT05623605
Title: Evaluation of Antibacterial Potency of New Different Herbal Mouthwashes Against Caries Forming Bacteria, a Randomized Control Trial
Brief Title: Evaluation of New Different Herbal Mouthwashes Against Caries Forming Bacteria, RCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nahda University (Other)
Responsible Party: Principal Investigator, GHada Abdelwahab Ahmed, Associate Professor of Pediatric Dentistry, Nahda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 040522
Record Dates: First submitted 2022-11-12; First posted 2022-11-21 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Dental Caries in Children
Keywords: Moringa; Star Anis; Indian Costus; Mouth wash; Streptococus Mutans

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moringa mouthwash (Experimental): 5 ml Moringa mouthwash two times per day for 1 week
  Interventions: Drug: Moringa mouthwash
- Star Anis mouthwash (Experimental): 5 ml Star Anis mouthwash two times per day for 1 week
  Interventions: Drug: star anise mouthwash
- Indian Costus mouthwash (Experimental): 5 ml Indian Costus mouthwash two times per day for 1 week
  Interventions: Drug: Indian costus mouth wash

INTERVENTIONS:
Drug: Moringa mouthwash — using Moringa mouthwashes in 3 different concentrations (5,10,15%) twice per day for 7 days
  Other Names: Moringa herbal mouthwash
  Arms: Moringa mouthwash
Drug: star anise mouthwash — using star anise mouthwash in 3 different concentrations (5,10,15%) twice per day for 7 days
  Other Names: star anise herbal mouthwash
  Arms: Star Anis mouthwash
Drug: Indian costus mouth wash — using Indian costus mouthwash in 3 different concentrations (5,10,15%) twice per day for 7 days
  Other Names: Indian costus herbal mouth wash
  Arms: Indian Costus mouthwash

SUMMARY:
The goal of this randomized controlled trial is to compare three different types of mouthwash, Moringa, Star anis, and Indian Costus 90 children participated in this study divided into 3 groups according to the type of mouthwash used and then subdivided in each group into 3 subgroups according to the concentration of the mouthwash 5,10,15%. the children were asked to rinse with the mouthwash 3 times per day for 1 week. bacterial count for streptococcus mutans was measured before and after the use of mouthwash to see the most effective concentration.

DETAILED DESCRIPTION:
The powdered of Moringa, Star anis, and Indian Costus leaves (250 g) were extracted using 90% ethanol then filtered using Whatman Filter paper No.1 and dried under reduced pressure using rota vapor. The crude ethanolic extract was (200 mg). ninety children will be randomly distributed into three groups (1,2,3) (30 children each). each group was divided into further 3 groups (10 children each) according to the concentration of each herbal mouthwash (5,10,15%). each participant will be given a new bottle of a specific effective amount of herbal extract to be used as a mouthwash. Children will be instructed to rinse with 5ml of mouthwash. All groups were instructed to rinse three times a day with specific mouthwash for each group for about one minute and participants will be advised to use the mouthwash for seven days. Collection of saliva samples Prior to the start of the experiment, samples of unstimulated saliva were taken when the child spit a suitable amount of unstimulated saliva in a sterile container in the morning before breakfast. Initial salivary samples were collected to establish base levels (S1) using selective culture media, The salivary samples (S2) were collected after one week of using the mouthwash when the child spit a suitable amount of unstimulated saliva in a sterile container in the morning before breakfast.

ELIGIBILITY:
Inclusion Criteria:

* - Children with no systemic disease, no history of recent antibiotic administration (last 2 weeks), antimicrobial mouth-rinse (last 12 hours), topical fluoride treatment within 4 weeks prior to baseline, children with no untreated active carious lesion, no orthodontic appliance or with low caries index (DMF& def < 4)

Exclusion Criteria:

* Children using antibiotics, medications or mouthwashes at the time of the study, children with oral or systemic disease, children undergoing any dental treatment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-06-19 (Actual); Primary Completion 2022-12-13 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
bacterial count | 1 weak
  decrease the count of streptococus mutans after use of the herbal mouthwash

CONTACTS AND LOCATIONS:
Overall Officials: Mariem Elmansy, Ph.D, Study Chair — researcher
Locations (1):
- Ghada Salem, Maadi, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No